CLINICAL TRIAL: NCT04321226
Title: Femtosecond Laser-assisted Astigmatism Treatment (FLAAT)
Brief Title: Femtosecond Laser-assisted Astigmatism Treatment
Acronym: FLAAT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Rupert Menapace, Clinical Professor, Medical University of Vienna
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1422/2017
Record Dates: First submitted 2020-03-23; First posted 2020-03-25 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Age Related Cataracts; Astigmatism
Keywords: Laser Cataract Surgery; Arcuate Keratotomy
MeSH Terms: conditions — Astigmatism

STUDY DESIGN:
Intervention Model Description: Prospective interventional case series
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Femtosecond Laser guided Arcuate Keratotomy (Experimental): Arcuate keratotomy will be performed together with Laser cataract surgery
  Interventions: Device: Femtosecond Laser guided Arcuate Keratotomy

INTERVENTIONS:
Device: Femtosecond Laser guided Arcuate Keratotomy — Astigmatism will be reduced in cataract surgery using a low energy Femtosecond Laser device

SUMMARY:
The investigational device is an approved femtosecond laser (FSL) device with an integrated imaging system to perform certain steps of the cataract procedure including arcuate incisions (AI) correcting astigmatism, also referred to as arcuate keratotomy (AK). The FSL will perform anterior capsulotomy and lens fragmentation in individuals suffering from age-related cataract with need of cataract surgery and additionally perform arcuate keratotomy in individuals with more than 1.0 Diopter (dpt) of astigmatism. Cataract surgery will be performed in subjects who have signed an informed consent form.

Postoperative examinations will be implemented in accordance with the approved Investigational Plan on subjects and includes: postoperative refraction, visual acuity, slitlamp examination, and corneal topography

ELIGIBILITY:
Inclusion Criteria:

* Age-related cataract necessitating lens extraction and posterior IOL implantation
* Regular corneal astigmatism between 1.0 and 2.5 DPT
* Age 40 and older (females of childbearing age will be interviewed if pregnancy is possible)

Exclusion Criteria:

* Corneal abnormality
* Preceding ocular surgery or trauma
* Uncontrolled glaucoma
* Proliferative diabetic retinopathy
* Iris neovascularization
* History of uveitis/iritis
* Microphthalmus
* Recurrent intraocular inflammation of unknown etiology
* Blind fellow eye
* Uncontrolled systemic or ocular disease

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2017-07-10 (Actual); Primary Completion 2022-03-05 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
Corneal Astigmatism one year after the intervention | 1 year follow-up
  H0: no change in postoperative refraction astigmatism H1: change in postoperative refraction astigmatism

SECONDARY OUTCOMES:
Precision and reproducibility of corneal cut depth | 1 year follow-up
  Corneal Incisions will be measured using an anterior segment SS-OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria